CLINICAL TRIAL: NCT05700344
Title: Multicentric, Observational Study to Evaluate Real World Data of Avelumab in First Line Maintenance Therapy for Advanced or Metastatic Urothelial Carcinoma, a SOGUG Study
Brief Title: SOGUG-AVELUMAB_RWD
Acronym: SOGUG
Status: Completed | Type: Observational
Sponsor: Spanish Oncology Genito-Urinary Group (Other)
Collaborators: Adknoma Health Research (Industry)
Responsible Party: Sponsor
Other Study IDs: SOGUG-2021-IEC(VEJ)-5
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — avelumab

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Avelumab — Single Group Assignment

SUMMARY:
The study goal is to evaluate the effectiveness in clinical practice of Avelumab as first line maintenance therapy in patients with locally advanced or metastatic Urothelial Carcinoma, who have not progressed after first line platinum-based treatment.

Study is performed at national hospitals from approximately 22 different sites and expecting to recruit 120 patients.

Patients understanding the nature of the study by providing their informed consent prior to participation.

* Patients of both sexes diagnosed with locally advanced or metastatic Urothelial Carcinoma, stage IV disease before first line with carboplatin/cisplatin-based chemotherapy. No disease progression after four-six cycles of ChT according to the Response Evaluation Criteria in Solid Tumor with a treatment free interval of 4-10 weeks before Avelumab initiation date.
* Patients who started Avelumab as maintenance therapy in first line after 21/Jan./2021 and before 27/Apr./2022 (both dates included).

DETAILED DESCRIPTION:
Multicentre, observational, ambispective (retrospective and prospective) study to evaluate the real-world evidence of Avelumab as maintenance therapy in patients diagnosed with Urothelial Carcinoma (WHO classification) and previously treated with platinum-based treatment in first line. Study is performed at national hospitals from approximately 22 different sites and expecting to recruit 120 patients. Patients are selected based on the existing medical record of have been treated with Avelumab as maintenance therapy in first line before initiating the study (retrospective data); patients who continues receiving Avelumab after inclusion will also contribute to data collection until the end of treatment or end of study (prospective data).

According to mUC incidence and the selective inclusion criteria from this study of having initiated Avelumab as maintenance therapy in 1L between EMA approval date (Jan. 2021) and date of national reimbursement prize (Apr.2022), which is a narrow period of time to recruit the necessary number of candidates, therefore, prospective data from each participant patient will be a key to ensure the assessment of the study objective eventually.

Investigators will review the medical history of patients treated or under treatment of Avelumab and select chronologically those who matches the inclusion criteria. Patients will be informed during a regular follow up visit about the nature of the study and requested to sign the patient consent form once the decision of participating is made. At this point, the retrospective data from patients is collected (such as demographics, toxicity, anthropometrics, vital signs, comorbidities, hemogram, dosage modification etc.) previous adverse reactions (ARs) and serious adverse reaction (SARs) related to Avelumab. Included patients, that continues under Avelumab treatment will be monitored by investigators and prospective data from them will be collected during follow up visits and/or from electronic medical records (eMR).

Deceased patient who fulfils the inclusion criteria can be also included, being able to access to its clinical data at the beginning of the study according to Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data, and repealing Directive 95/46/EC (General Data Protection Regulation) and the Spanish Organic Law 3/2018 of 5th December, on the protection of personal data and digital rights. Additionally, the investigator team will consult in the eMR of deceased patients to ensure that they did not express in life opposition to the use of their data for investigational purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients understanding the nature of the study by providing their informed consent prior to participation.
* Patients of both sexes diagnosed with locally advanced or metastatic Urothelial Carcinoma, stage IV disease (AJCC ed. 8th, 2017) before first line with carboplatin/cisplatin-based chemotherapy (ChT). No disease progression after four-six cycles of ChT according to the Response Evaluation Criteria in Solid Tumor (RECIST 1.1) with a treatment free interval of 4-10 weeks before Avelumab initiation date.
* Patients who started Avelumab as maintenance therapy in first line after 21/Jan./2021 and before 27/Apr./2022 (both dates included).

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with locally advanced or metastatic Urothelial Carcinoma who have not progressed after first line platinum-based treatment and who received or are receiving Avelumab as the first-line maintenance therapy in routine clinical practice.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-11-02 (Actual)

PRIMARY OUTCOMES:
Median progression free survival (mPFS) | Throughout the study period. Approximately 8 months
  median time for patients from treatment initiation with Bavencio® to the date of real world progression event or death due to any cause. Patients without a real-world progression event or date of death will be censored at the most recent visit with the treating oncologist or end of follow up.

SECONDARY OUTCOMES:
Median overall survival (mOS) | Throughout the study period. Approximately 8 months
  median length of the time from the date patient initiates treatment with Bavencio® to the date of death. Patients not dead will be censored at the most recent visit with the treating oncologist or end of follow up.
Progression free survival rate at 12 months (PFS12) | Throughout the study period. Approximately 8 months
  percentage of alive patients and progression free 12 month after treatment initiation with Bavencio®. Patients without a real-world progression event or date of death will be censored at month 12th.
Collection of any adverse reaction (AR) or serious adverse reaction (SAR) | Throughout the study period. Approximately 8 months
  Collection of any adverse reaction (AR) or serious adverse reaction (SAR) occurring during treatment period (retrospective and prospective).
Collection of any adverse event (AE) or serious adverse event (SAE) | Throughout the study period. Approximately 8 months
  Collection of any adverse event (AE) or serious adverse event (SAE) during prospective data collection. Immune check points inhibitors have unique side effects known as immune-related adverse event (irAE) that along with the treatment related AE (TRAE) are of interest to the study (3, 4).

CONTACTS AND LOCATIONS:
Overall Officials: Áurea Molina, Principal Investigator — Complejo Hospitalario Universitario A Coruña (CHUAC); Ovidio Fernández, Principal Investigator — Complejo Hospitalario Universitario Ourense (CHOU)
Locations (22):
- Spain (22):
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Complejo Hospitalario Universitario Albacete, Albacete
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital Universitario Basurto, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - Hospital Provincial de Castellón, Castellon
  - Hospital Universitario Vinalopó, Elche
  - Hospital General Universitario de Elda, Elda
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Complexo Hospitalario Universitario Ourense, Ourense
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Río Carrión, Palencia
  - Hospital Sagunto, Sagunto
  - Hospital Universitario de Salamanca, Salamanca
  - Complexo Hospitalario Universitario Santiago, Santiago de Compostela
  - Fundación Instituto Valenciano de Oncología, Valencia
  - Hospital Universitario Politècnic La Fe, Valencia
  - Hospital Marina Baixa Villajosyosa, Villajoyosa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar V, Chaudhary N, Garg M, Floudas CS, Soni P, Chandra AB. Current Diagnosis and Management of Immune Related Adverse Events (irAEs) Induced by Immune Checkpoint Inhibitor Therapy. Front Pharmacol. 2017 Feb 8;8:49. doi: 10.3389/fphar.2017.00049. eCollection 2017. PMID 28228726
- [Background] Galsky MD, Balar AV, Black PC, Campbell MT, Dykstra GS, Grivas P, Gupta S, Hoimes CJ, Lopez LP, Meeks JJ, Plimack ER, Rosenberg JE, Shore N, Steinberg GD, Kamat AM. Society for Immunotherapy of Cancer (SITC) clinical practice guideline on immunotherapy for the treatment of urothelial cancer. J Immunother Cancer. 2021 Jul;9(7):e002552. doi: 10.1136/jitc-2021-002552. PMID 34266883
- [Background] Kim JW, Tomita Y, Trepel J, Apolo AB. Emerging immunotherapies for bladder cancer. Curr Opin Oncol. 2015 May;27(3):191-200. doi: 10.1097/CCO.0000000000000177. PMID 25811346
- [Background] Morales-Barrera R, Suarez C, Gonzalez M, Valverde C, Serra E, Mateo J, Raventos C, Maldonado X, Morote J, Carles J. The future of bladder cancer therapy: Optimizing the inhibition of the fibroblast growth factor receptor. Cancer Treat Rev. 2020 Jun;86:102000. doi: 10.1016/j.ctrv.2020.102000. Epub 2020 Mar 13. PMID 32203842
- [Background] Wolacewicz M, Hrynkiewicz R, Grywalska E, Suchojad T, Leksowski T, Rolinski J, Niedzwiedzka-Rystwej P. Immunotherapy in Bladder Cancer: Current Methods and Future Perspectives. Cancers (Basel). 2020 May 7;12(5):1181. doi: 10.3390/cancers12051181. PMID 32392774
- [Background] Powles T, Rosenberg JE, Sonpavde GP, Loriot Y, Duran I, Lee JL, Matsubara N, Vulsteke C, Castellano D, Wu C, Campbell M, Matsangou M, Petrylak DP. Enfortumab Vedotin in Previously Treated Advanced Urothelial Carcinoma. N Engl J Med. 2021 Mar 25;384(12):1125-1135. doi: 10.1056/NEJMoa2035807. Epub 2021 Feb 12. PMID 33577729
- [Background] Balar AV, Galsky MD, Rosenberg JE, Powles T, Petrylak DP, Bellmunt J, Loriot Y, Necchi A, Hoffman-Censits J, Perez-Gracia JL, Dawson NA, van der Heijden MS, Dreicer R, Srinivas S, Retz MM, Joseph RW, Drakaki A, Vaishampayan UN, Sridhar SS, Quinn DI, Duran I, Shaffer DR, Eigl BJ, Grivas PD, Yu EY, Li S, Kadel EE 3rd, Boyd Z, Bourgon R, Hegde PS, Mariathasan S, Thastrom A, Abidoye OO, Fine GD, Bajorin DF; IMvigor210 Study Group. Atezolizumab as first-line treatment in cisplatin-ineligible patients with locally advanced and metastatic urothelial carcinoma: a single-arm, multicentre, phase 2 trial. Lancet. 2017 Jan 7;389(10064):67-76. doi: 10.1016/S0140-6736(16)32455-2. Epub 2016 Dec 8. PMID 27939400
- [Background] Balar AV, Castellano D, O'Donnell PH, Grivas P, Vuky J, Powles T, Plimack ER, Hahn NM, de Wit R, Pang L, Savage MJ, Perini RF, Keefe SM, Bajorin D, Bellmunt J. First-line pembrolizumab in cisplatin-ineligible patients with locally advanced and unresectable or metastatic urothelial cancer (KEYNOTE-052): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2017 Nov;18(11):1483-1492. doi: 10.1016/S1470-2045(17)30616-2. Epub 2017 Sep 26. PMID 28967485
- [Background] Sharma P, Retz M, Siefker-Radtke A, Baron A, Necchi A, Bedke J, Plimack ER, Vaena D, Grimm MO, Bracarda S, Arranz JA, Pal S, Ohyama C, Saci A, Qu X, Lambert A, Krishnan S, Azrilevich A, Galsky MD. Nivolumab in metastatic urothelial carcinoma after platinum therapy (CheckMate 275): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2017 Mar;18(3):312-322. doi: 10.1016/S1470-2045(17)30065-7. Epub 2017 Jan 26. PMID 28131785
- [Background] Bukhari N, Al-Shamsi HO, Azam F. Update on the Treatment of Metastatic Urothelial Carcinoma. ScientificWorldJournal. 2018 Jun 6;2018:5682078. doi: 10.1155/2018/5682078. eCollection 2018. PMID 29977169
- [Background] von der Maase H, Sengelov L, Roberts JT, Ricci S, Dogliotti L, Oliver T, Moore MJ, Zimmermann A, Arning M. Long-term survival results of a randomized trial comparing gemcitabine plus cisplatin, with methotrexate, vinblastine, doxorubicin, plus cisplatin in patients with bladder cancer. J Clin Oncol. 2005 Jul 20;23(21):4602-8. doi: 10.1200/JCO.2005.07.757. PMID 16034041
- [Background] von der Maase H, Hansen SW, Roberts JT, Dogliotti L, Oliver T, Moore MJ, Bodrogi I, Albers P, Knuth A, Lippert CM, Kerbrat P, Sanchez Rovira P, Wersall P, Cleall SP, Roychowdhury DF, Tomlin I, Visseren-Grul CM, Conte PF. Gemcitabine and cisplatin versus methotrexate, vinblastine, doxorubicin, and cisplatin in advanced or metastatic bladder cancer: results of a large, randomized, multinational, multicenter, phase III study. J Clin Oncol. 2000 Sep;18(17):3068-77. doi: 10.1200/JCO.2000.18.17.3068. PMID 11001674
- [Background] Grivas P, Agarwal N, Pal S, Kalebasty AR, Sridhar SS, Smith J, Devgan G, Sternberg CN, Bellmunt J. Avelumab first-line maintenance in locally advanced or metastatic urothelial carcinoma: Applying clinical trial findings to clinical practice. Cancer Treat Rev. 2021 Jun;97:102187. doi: 10.1016/j.ctrv.2021.102187. Epub 2021 Mar 22. PMID 33839438
- [Background] Apolo AB, Infante JR, Balmanoukian A, Patel MR, Wang D, Kelly K, Mega AE, Britten CD, Ravaud A, Mita AC, Safran H, Stinchcombe TE, Srdanov M, Gelb AB, Schlichting M, Chin K, Gulley JL. Avelumab, an Anti-Programmed Death-Ligand 1 Antibody, In Patients With Refractory Metastatic Urothelial Carcinoma: Results From a Multicenter, Phase Ib Study. J Clin Oncol. 2017 Jul 1;35(19):2117-2124. doi: 10.1200/JCO.2016.71.6795. Epub 2017 Apr 4. PMID 28375787
- [Background] O'Donnell JC, Le TK, Dobrin R, Higashi M, Pereira A, Wagner S, Yang A, Hukkelhoven M. Evolving use of real-world evidence in the regulatory process: a focus on immuno-oncology treatment and outcomes. Future Oncol. 2021 Jan;17(3):333-347. doi: 10.2217/fon-2020-0591. Epub 2020 Oct 19. PMID 33074018
- [Background] Cramer-van der Welle CM, Verschueren MV, Tonn M, Peters BJM, Schramel FMNH, Klungel OH, Groen HJM, van de Garde EMW; Santeon NSCLC Study Group. Real-world outcomes versus clinical trial results of immunotherapy in stage IV non-small cell lung cancer (NSCLC) in the Netherlands. Sci Rep. 2021 Mar 18;11(1):6306. doi: 10.1038/s41598-021-85696-3. PMID 33737641
- [Background] Pasello G, Pavan A, Attili I, Bortolami A, Bonanno L, Menis J, Conte P, Guarneri V. Real world data in the era of Immune Checkpoint Inhibitors (ICIs): Increasing evidence and future applications in lung cancer. Cancer Treat Rev. 2020 Jul;87:102031. doi: 10.1016/j.ctrv.2020.102031. Epub 2020 May 16. PMID 32446182
- [Background] Stewart M, Norden AD, Dreyer N, Henk HJ, Abernethy AP, Chrischilles E, Kushi L, Mansfield AS, Khozin S, Sharon E, Arunajadai S, Carnahan R, Christian JB, Miksad RA, Sakoda LC, Torres AZ, Valice E, Allen J. An Exploratory Analysis of Real-World End Points for Assessing Outcomes Among Immunotherapy-Treated Patients With Advanced Non-Small-Cell Lung Cancer. JCO Clin Cancer Inform. 2019 Jul;3:1-15. doi: 10.1200/CCI.18.00155. PMID 31335166
- [Background] Aly A, Johnson C, Yang S, Botteman MF, Rao S, Hussain A. Overall survival, costs, and healthcare resource use by line of therapy in Medicare patients with newly diagnosed metastatic urothelial carcinoma. J Med Econ. 2019 Jul;22(7):662-670. doi: 10.1080/13696998.2019.1591424. Epub 2019 Mar 25. PMID 30836812
- [Result] Powles T, Park SH, Voog E, Caserta C, Valderrama BP, Gurney H, Kalofonos H, Radulovic S, Demey W, Ullen A, Loriot Y, Sridhar SS, Tsuchiya N, Kopyltsov E, Sternberg CN, Bellmunt J, Aragon-Ching JB, Petrylak DP, Laliberte R, Wang J, Huang B, Davis C, Fowst C, Costa N, Blake-Haskins JA, di Pietro A, Grivas P. Avelumab Maintenance Therapy for Advanced or Metastatic Urothelial Carcinoma. N Engl J Med. 2020 Sep 24;383(13):1218-1230. doi: 10.1056/NEJMoa2002788. Epub 2020 Sep 18. PMID 32945632
- See also: ASC. American Cancer Society. Bladder cancer — https://www.cancer.org/cancer/bladder-cancer/about.html
- Available data/document: Summary of Product Characteristics — https://www.ema.europa.eu/en/documents/product-information/bavencio-epar-product-information_en.pdf — Summary of Product Characteristics
- Available data/document: Burki TK. Erdafitinib for advanced urothelial carcinoma — http://dx.doi.org/10.1016/S1470-2045(19)30522-4 — Burki TK. Erdafitinib for advanced urothelial carcinoma. Lancet Oncology Vol.20 September 2019. Published Online August 1, 2019